CLINICAL TRIAL: NCT01081093
Title: Biventricular Pacing in Hypertrophic Cardiomyopathy After Aortic Valve Replacement
Acronym: BIVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, PI, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bivent001AR-AHK
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic Cardiomyopathy Diastolic Ventricular Interaction; Biventricular Pacemaker cardiac surgery aortic valve replacement
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biventricular pacing (Experimental)
  Interventions: Procedure: additional temporary pacewire

INTERVENTIONS:
Procedure: additional temporary pacewire — Placement of an additional pacing wire on the left side of the heart after aortic valve replacement in patients with hypertrophic cardiomyopathy

SUMMARY:
Biventricular Pacing has been shown an improvement of symptoms in patients with heart failure.

A temporary pacing is necessary in patients after cardiac procedures. In patients with hypertrophic cardiomyopathy, a single right ventricular pacing can decrease the cardiac output and blood pressure.

The investigators propose that biventricular pacing in these patients and conditions results in an improvement of symptoms instead of single right pacing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Hypertrophic Cardiomyopathy
* Aortic valve replacement

Exclusion Criteria:

* Atrial fibrillation
* Pericarditis
* postoperative low output
* Preoperative permanent pacemaker placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Cardiac output | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe Universitätsklinikum, Frankfurt am Main, Germany